CLINICAL TRIAL: NCT04698980
Title: Evaluation of the STANDARD G6PD Rapid Test for Assaying the Enzymatic Activity of G6PD in French Guiana
Acronym: G6PD facile
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut Pasteur de la Guyane (Unknown); Centre Hospitalier Andrée Rosemon de Cayenne (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-015
Record Dates: First submitted 2020-12-18; First posted 2021-01-07 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Paludism
Keywords: paludism; French Guiana; G6PD; rapid diagnostic test; STANDARD G6PD
MeSH Terms: conditions — Malaria | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: 150 participants selected according to their G6PD activity:
  * 50 subjects with "severe deficit" G6PD activity (<30% of the median in the general population, ie 3.6U / g Hb), adults or children two years and over.
  * 50 subjects with "intermediate" G6PD activity (30-80%), adults.
  * 50 subjects with "normal" G6PD activity (> 80% ie> 9.6U / g Hb), adults.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants selected according to their G6PD activity (Other): * 50 subjects with "severe deficit" G6PD activity (<30% of the median in the general population, ie 3.6U / g Hb), adults or children two years and over.
  * 50 subjects with "intermediate" G6PD activity (30-80%), adults.
  * 50 subjects with "normal" G6PD activity (> 80% ie> 9.6U / g Hb), adults.
  Interventions: Diagnostic Test: blood samples (venous and capillary at the fingertip)

INTERVENTIONS:
Diagnostic Test: blood samples (venous and capillary at the fingertip) — For each participant, the intervention will be a fingertip sample to perform the STANDARD G6PD test and two blood samples on EDTA to perform the reference test

SUMMARY:
In French Guiana, malaria is endemic and two species predominate: P. falciparum and P. vivax. The treatments against Plasmodium vivax malaria are: nivaquine for 3 days against circulating blood parasites and primaquine for 14 days against parasites dormant in the liver. Primaquine can cause iatrogenic hemolytic anemias in patients with favism, i.e. G6PD deficiency. This anemia can be severe enough to cause the death of the deficient patient. Thus, the WHO and HCSP recommendations indicate that a quantitative assay of the activity of this enzyme should be carried out before its prescription. This deficiency is a recessive inherited disease linked to the X chromosome characterized by more or less low levels of enzymatic activity which depends on the genotype of the patients but not only because the phenotype depends on the level of activation of the X chromosome for each cell.

Currently, obtaining a G6PD assay in French Guiana is a long process since it is done in mainland France and the pre-analytical conditions are quite demanding. Thus, in areas of transmission of P. vivax, patients usually have a bout of revival before being prescribed primaquine. This period includes: dosing G6PD at a distance from access, obtaining the result and then the nominal ATU to finally obtain and deliver the primaquine.

DETAILED DESCRIPTION:
This is a interventional,prospective, multicenter, cross-sectional and comparative study.

To achieve this study, the following will be done:

* Selection of subjects according to their G6PD activity from the list of participants previously included in the ELIMALAR Palustop study and from known LHUPM patients in Cayenne following a request for a G6PD dosage, whether or not related to malaria.
* Collection of clinical data from participants (sex, age, ethnicity of parents and grandparents).
* Collection of blood samples from subjects showing G6PD activity of the following three categories "severe deficiency", "intermediate", "normal".
* Determination of G6PD activity by the "STANDARD G6PD" technique from SD BIOSENSOR versus the reference enzymatic method

ELIGIBILITY:
Inclusion Criteria:

* People with a known level of G6PD activity.
* People or their legal representatives who have received information on the research and have signed a written consent to participate in the study
* People aged over 18 for the "intermediate" and "normal" categories,
* People aged two years and over for the "severe deficit" category.

Exclusion Criteria:

* People with an unknown level of G6PD activity,
* People or their legal representatives who refused to participate in the study,
* People aged under 18 for the intermediate and normal categories,
* Children under 2 years old for the "severe deficit" category,
* People with a hemoglobin level below 11g / dL for men and 10g / dL for women and children.
* People who received a transfusion less than 4 months before the proposal to participate in the G6PD study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the STANDARD G6PD test | 3 years
  The sensitivity and specificity will be calculated for the detection of severe deficits in G6PD activity (<30%), intermediate activities (30-80%) and normal activities (> 80%) of the STANDARD G6PD test vs the reference enzymatic method

SECONDARY OUTCOMES:
Verification of the analysis method by the STANDARD G6PD test several times | 3 years
  Measurement of the G6PD activity will be done to assess the repeatability, accuracy or trueness of the STANDARD G6PD test according to the recommendations of standard NF EN ISO 15189: 2012 for accreditation.
Verification of the analysis method by the STANDARD G6PD test by different operator | 3 years
  Measurement of the G6PD activity will be done to assess the inter-operator variability, of the STANDARD G6PD test according to the recommendations of standard NF EN ISO 15189: 2012 for accreditation.
Verification of the analysis method by the STANDARD G6PD test in different conditions | 3 years
  Measurement of the G6PD activity will be done to assess the reproducibility, robustness and measurement interval of the STANDARD G6PD test according to the recommendations of standard NF EN ISO 15189: 2012 for accreditation.
sequencing of the coding regions of the G6PD gene of 150 individuals | 3 years
  Analysis of the genotype of the G6PD gene and comparison to the phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Lise Musset, PharmD, Principal Investigator — Institut Pasteur de la Guyane, head of Parasitology laboratory
Locations (1):
- Institut Pasteur de la Guyane, Cayenne, French Guiana